CLINICAL TRIAL: NCT03916198
Title: Effect of Polydeoxyribonucleotide (PDRN) on Healing and Fatty Degeneration of Rotator Cuff in Human
Brief Title: Polydeoxyribonucleotide (PDRN) for Cuff Regeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Associate Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-01-021
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Tear
Keywords: healing; fatty degeneration; retear
MeSH Terms: conditions — Rotator Cuff Injuries; Fatty Liver | interventions — Polydeoxyribonucleotides; Saline Solution

STUDY DESIGN:
Intervention Model Description: 79 participants with rotator cuff tear will be classified into two group. One group (PDRN) will be injected at the repaired cuff with 3cc polydeoxyribonucleotide just after surgery and be injected with another 3cc polydeoxyribonucleotide under ultrasound guidance 2 weeks after the surgery. The other group (CONTROL) will be injected with 3ml normal saline in the same manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 79 participants with rotator cuff tear will be randomly assigned to PDRN or CONTROL depending on the injection material. Randomization will be performed with a computerized random-sequence generator by an independent nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDRN(polydeoxyribonucleotide) (Experimental): polydeoxyribonucleotide 3cc at surgery under arthroscopy guidance and 2 weeks after surgery under ultrasound guidance
  Interventions: Drug: Polydeoxyribonucleotides
- CONTROL(normal saline) (Placebo Comparator): normal saline 3cc at surgery under arthroscopy guidance and 2 weeks after surgery under ultrasound guidance
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Polydeoxyribonucleotides — Just after arthroscopic rotator cuff repair, 3cc polydeoxyribonucleotide will be injected, and 2 weeks after the surgery the same amount of the material will be injected.
  Other Names: PDRN
  Arms: PDRN(polydeoxyribonucleotide)
Drug: Normal saline — Just after arthroscopic rotator cuff repair, 3cc normal saline will be injected, and 2 weeks after the surgery the same amount of the material will be injected.
  Arms: CONTROL(normal saline)

SUMMARY:
This study is to evaluate the effect of polydeoxyribonucleotide (PDRN) for healing and fatty degeneration of rotator cuff. The investigators will enroll 130 patients with rotator cuff tear who will undergo arthroscopic rotator cuff repair. 130 patients will be classified into two group. One group (PDRN) will be injected at the repaired cuff with 3cc polydeoxyribonucleotide just after surgery and be injected with another 3ml polydeoxyribonucleotide under ultrasound guidance 2 weeks after the surgery. The other group (CONTROL) will be injected with 3ml normal saline in the same manner.

DETAILED DESCRIPTION:
Polydeoxyribonucleotide is a tissue regeneration activator. It binds an adenosine receptor and stimulate VEGF(vascular endothelial growth factor) synthesis and stimulate collagen synthesis. Nowadays, a lot of arthroscopic rotator cuff repairs are being performed. but the failure rate of rotator cuff repair is considerably high. Therefore, this study is to evaluate the effect of polydeoxyribonucleotide for healing and fatty degeneration of rotator cuff.

Visual analog scale (VAS) of pain and other functional scores of the two group will be checked preoperatively and postoperative 3, 6, 12, 24 months. Growth factors (VEGF, fibroblast growth factor(FGF), insulin like growth factor(IGF)) will be checked preoperatively and postoperative 1h, 2 days, 2 weeks, 6 weeks, 3, 6 months. Follow up MRI will be checked at postoperative 6 months. The parameters will be compared using statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* definite rotator cuff tear on preoperative MRI, which needs repair
* acceptance of arthroscopic surgery including rotator cuff repair

Exclusion Criteria:

* history of ipsilateral shoulder operation or fracture
* concomitant neurological disorder around the

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow score | 2 years
  functional score of shoulder between 0 to 100(0: bad, 100: good)

SECONDARY OUTCOMES:
Constant score | 2 years
  functional score of shoulder between 0 to 100(0: bad, 100: good)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD,PhD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is a privacy problem. The investigators should negotiate with our government about that.

REFERENCES:
- [Background] Altavilla D, Squadrito F, Polito F, Irrera N, Calo M, Lo Cascio P, Galeano M, La Cava L, Minutoli L, Marini H, Bitto A. Activation of adenosine A2A receptors restores the altered cell-cycle machinery during impaired wound healing in genetically diabetic mice. Surgery. 2011 Feb;149(2):253-61. doi: 10.1016/j.surg.2010.04.024. Epub 2010 Jun 8. PMID 20570301
- [Background] Galeano M, Bitto A, Altavilla D, Minutoli L, Polito F, Calo M, Lo Cascio P, Stagno d'Alcontres F, Squadrito F. Polydeoxyribonucleotide stimulates angiogenesis and wound healing in the genetically diabetic mouse. Wound Repair Regen. 2008 Mar-Apr;16(2):208-17. doi: 10.1111/j.1524-475X.2008.00361.x. PMID 18318806
- [Result] Kang SH, Choi MS, Kim HK, Kim WS, Bae TH, Kim MK, Chang SH. Polydeoxyribonucleotide improves tendon healing following achilles tendon injury in rats. J Orthop Res. 2018 Jun;36(6):1767-1776. doi: 10.1002/jor.23796. Epub 2017 Nov 28. PMID 29094396

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT03916198/Prot_SAP_000.pdf